CLINICAL TRIAL: NCT05640128
Title: Determination of Threshold Values of Aldosterone in HPLC-MS/MS, of Renin and of the Aldosterone / Renin Ratio for the Diagnosis of Primary Hyperaldosteronism
Acronym: DAPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-209
Record Dates: First submitted 2022-11-28; First posted 2022-12-07 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-11

CONDITIONS: Hyperaldosteronism; Primary
MeSH Terms: conditions — Hyperaldosteronism | interventions — Aldosterone; Liquid Chromatography-Mass Spectrometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aldosterone in HPLC-MS/MS, (Other): Aldosterone in HPLC-MS/MS measurement
  Interventions: Other: Aldosterone in HPLC-MS/MS

INTERVENTIONS:
Other: Aldosterone in HPLC-MS/MS — Aldosterone in HPLC-MS/MS

SUMMARY:
collaborative work within 2 hospitals at the CHU of Caen, at the CHRU of Lille, concerning the evaluation of the biological markers of primary hyperaldosteronism (PAH) with the dosage of aldosterone in LC -MS/MS, which is performed in both centers, with two different techniques. The main objective is to define the range of Aldosterone concentrations in LC MS/MS, of renin in an automated method, in populations of healthy volunteers, essential hypertensives, and hypertensives with primary hyperaldosteronism. , in order to establish a threshold for the screening of PAH by the RAR, and for the confirmation of PAH by a dynamic test with an Aldosterone threshold post salt load test.

ELIGIBILITY:
Inclusion Criteria:

* Patients (18-75 years old) with moderate to severe hypertension, which justifies carrying out an etiological assessment in a hospital environment.
* Assessment carried out in compliance with the standardized measurement conditions of the RAR defined by the SFE consensus,
* Signature of a written consent by the patient

Exclusion Criteria:

* Patient on antihypertensive treatment other than alpha-blockers, calcium channel blockers or centrally acting antihypertensive
* Etiology of secondary hypertension other than PAH

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-01-02 (Actual); Primary Completion 2023-01-02 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Aldosterone values in LC-MS/MS (and renin) and RAR calculation and calculation of an RAR threshold for PAH screening which differentiates between essential hypertension and PAH. | baseline
  Define the range of concentrations of Aldosterone in LC MS/MS, of renin in an automated immunological method with calculation of the RAR, in populations of healthy volunteers, essential hypertensives, and hypertensives with primary hyperaldosteronism , in order to establish a threshold for the detection of PAH by the RAR, and for the confirmation of PAH by a dynamic test of confirmation by Aldosterone.

CONTACTS AND LOCATIONS:
Locations (1):
- CAEN University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No